CLINICAL TRIAL: NCT05874518
Title: Clinical Observation of Warm Needling Combined With and Electroacupuncture Therapy on Ovulatory Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liuzhou Maternity and Child Healthcare Hospital (Other)
Responsible Party: Principal Investigator, Fanghua Yang, Director, Liuzhou Maternity and Child Healthcare Hospital
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: LiuzhouMCHH
Record Dates: First submitted 2023-04-11; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Warm Needling; Electroacupuncture; Ovulation Dysfunction
MeSH Terms: interventions — Electroacupuncture; Letrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Ask the patient to empty the bladder, and take supine position. Take guanyuan, zhongji, bilateral Tianshu, zigong, guilai, sanyinjiao, Taixi, zusanli, hegu points. Select 0.3mm×40mm fine needles. After conventional disinfection, the needle is 0.5-1 inch deep. Then the 1.5 cm moxa cones were inserted into the tail of the needle of the bilateral sanyinjioa and zusnli points for moxibustion. At the same time, electroacupuncture therapy was used. Select the density wave and set the time for 25 minutes.
  Generally, the patient feels comfortable as moderate, so that the patient feel acid, distension, heat or local muscles for rhythmic contraction. After treatment, first reduce the power to zero value, turn off the power supply, then remove the electrode clip from the needle handle, and pull out the fine needle stabbed into the tissue. Treatment begins on the 5th day of the menstrual cycle, qd (once a day), usually for 6-8 consecutive days, and continuing to the day of ovulation.
  Interventions: Other: warm needling combined with electroacupuncture
- Control group (Active Comparator): Treatment was started on day 5 of the menstrual cycle. Letrozole tablets were given at 2.5mg (Jiangsu Hengrui Pharmaceutical Co., Ltd., H19991001, 2.5mg per tablet), po (oral), qd, for 5-7 consecutive days. When the diameter of follicles reaches 18mm, Chorionic gonadotrophin is given at 5000u (Lizhu Group Lizhu Pharmaceutical Factory, Chinese medicine H44020668, 5000u per branch), with intramuscular injection, qd, to promote follicle discharge. Patients were also instructed to have sexual intercourse on the same day and on day 2.
  Interventions: Drug: The treatment with letrozole tablets was started on the fifth day of the menstrual cycle

INTERVENTIONS:
Other: warm needling combined with electroacupuncture — Treatment begins on the 5th day of the menstrual cycle, qd (once a day), usually for 6-8 consecutive days, and continuing to the day of ovulation.
  Arms: Experimental group
Drug: The treatment with letrozole tablets was started on the fifth day of the menstrual cycle — Letrozole tablets were given at 2.5mg (Jiangsu Hengrui Pharmaceutical Co., Ltd., H19991001, 2.5mg per tablet), po (oral), qd, for 5-7 consecutive days. When the diameter of follicles reaches 18mm, Chorionic gonadotrophin is given at 5000u (Lizhu Group Lizhu Pharmaceutical Factory, Chinese medicine H44020668, 5000u per branch), with intramuscular injection, qd, to promote follicle discharge. Patients were also instructed to have sexual intercourse on the same day and on day 2.
  Arms: Control group

SUMMARY:
To observe the effect of warm needling combined with electroacupuncture on the ovulation promotion rate and pregnancy rate in luteinized unruptured follicle syndrome (LUFS).

ELIGIBILITY:
Inclusion Criteria:

* Infertility diagnosis criteria refer to the "Obstetrics and Gynecology" [10]: Infertility refers to the patient fails to conceive a pregnancy with normal sexual life and without contraception for 1 year. In primary infertility, pregnancy has never occurred. In secondary infertility, patients have previously conceived, but are unable to conceive again without contraception for 1 year.
* The standard for ovulation infertility is formulated according to the first series of Guiding Principles for Clinical Research of New Chinese Medicine: Basal body temperature was continuously recorded for single phase for more than 3 months; Vaginal detached cell smear examination showed no significant periodic changes; Cervical mucus crystallization examination showed no periodic changes, and ellipsoid; There was no typical secretory period change in endometrial examination on 6 days before menstruation; a series of B-ultrasound monitoring showed no ovulation signs; Blood and urinary progesterone levels were lower than those in the luteal phase. Patients who met two of the above 6 items could be diagnosed with anovulation

Exclusion Criteria:

* Those who have any serious adverse reactions during the treatment process and cannot continue the treatment
* Failing to follow the treatment plan and receiving other treatment
* Patients who quit the treatment process by themselves, or who have an incomplete course of treatment, will have a negative effect on the curative effect

Ages: 23 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Ultrasound characteristics of ovulation | About 10 days on average until ≥18mm follicle disappears or 20mm follicle volume decreases
  Monitoring follicular intima thickness
vaginal B-ultrasound to monitor follicles (size and discharge) and endometrial thickness on the fifth day of menstruation | the endometrium of ≥8mm on the fifth day of menstruation
  vaginal B-ultrasound to monitor follicles (size and discharge) and endometrial thickness on the fifth day of menstruation
Use vaginal B-ultrasound to monitor follicles (size and discharge) and endometrial thickness on the fifth day of menstruation | 48 hours after chorionic gonadotropin injection
  When the follicle size reached 18mm and Chorionic gonadotrophin was injected
Pregnancy judgment | 14 days after ovulation
  Pregnancy was determined by detecting serum HCG (human chorionic gonadotropin) 14 days after ovulation
Pregnancy judgment | about 50 days of pregnancy
  At about 50 days of pregnancy, pregnancy sac or fetal heart beat through vaginal B ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Fanghua Yang, Liuchow, Guangxi, China